CLINICAL TRIAL: NCT03869905
Title: Aquamin®, a Multi-mineral Natural Product From Red Marine Algae, as an Adjuvant Intervention for Mild Ulcerative Colitis and Ulcerative Colitis in Remission
Brief Title: Aquamin® as an Adjuvant Intervention for Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Muhammad N Aslam, MD (Other)
Responsible Party: Sponsor-Investigator, Muhammad N Aslam, MD, Associate Research Scientist, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUM00156676
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Remission
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Aquamin; maltodextrin

STUDY DESIGN:
Intervention Model Description: This pilot study includes individuals with mild ulcerative colitis / ulcerative colitis in remission, and is a randomized, double-blind, placebo-controlled trial with two parallel treatment groups for the first 90 days. Subjects on placebo will be crossed over to Aquamin® after the halfway visit at day 90. Subjects on Aquamin® will continue their treatment until the end.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aquamin® (Experimental): To be taken for 180 days
  Interventions: Drug: Aquamin®
- Placebo first then Aquamin® (Placebo Comparator): Placebo: To be taken for the first 90 days. Aquamin®: To be taken for the last 90 days (after crossover)
  Interventions: Drug: Aquamin®; Drug: Placebo first then Aquamin®

INTERVENTIONS:
Drug: Aquamin® — 4 capsules per day; 2 to be taken in the morning and 2 in the evening (containing approximately 800 mg calcium/day)
  Other Names: Nutritional
Drug: Placebo first then Aquamin® — 4 capsules per day; 2 to be taken in the morning and 2 in the evening
  Other Names: Maltodextrin
  Arms: Placebo first then Aquamin®

SUMMARY:
The purpose of this study is to determine if Aquamin® works as a potential treatment to improve symptoms and if it will induce remission in patients with mild Ulcerative Colitis and extend remission in Ulcerative Colitis in remission.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis with confirmed diagnosis by histology and endoscopy AND in stable remission for 3 months or more without therapy or with maintenance therapy (except steroids and antibiotics for 3 months) OR having a mild disease.
* A negative pregnancy test

Exclusion Criteria:

* No history or diagnosis of any of the following conditions: Crohn's disease, bleeding disorders, gastrointestinal or colonic malignancy, Kidney disease, including kidney "stones" or hypercalcemia, Coagulopathy/hereditary hemorrhagic disorders/ or receiving therapeutic doses of Coumadin or heparin.
* Ingested certain medications (Calcium, Vitamin D, fiber supplements and Non-steroidal anti-inflammatory drugs - NSAIDs) within 30 days of study start.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in ulcerative colitis clinical features / presentation as measured by the Inflammatory Bowel Disease Questionnaire (IBDQ) score | Up to day 180
  This is a self-administered questionnaire. There are 32 quality of life questions related to bowel function. Each response corresponds to a letter 'a' through 'g'. Whereas 'a' indicates high frequency and 'g' indicates minimal frequency. The total IBDQ score ranges between 32 and 224, with higher scores indicating better quality of life.
Change in clinical assessment /gastroenterologist's endoscopic findings based on Ulcerative Colitis Disease Activity Index (UCDAI)/Mayo Scoring | Up to day 180
  UCDAI/Mayo Scoring consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0= normal condition and 3 = severe disease condition. The total Mayo score ranges from 0 to 12, with higher scores indicating more severe disease.
Change in Cytokine levels of the colon tissue as measured by Interleukin 8 (IL-8) levels assessed by enzyme-linked immunosorbent assay (ELISA) | Up to day 180
  Interleukin 8 levels are measured in picograms per milliliter (pg/mL)
Change in serum C-reactive protein (CRP) levels as measured in a blood sample. | Up to day 180
  Serum C-reactive protein ([CRP levels)] will be reported in milligram per deciliter (mg/dL)
Change in fecal calprotectin levels measured in a stool sample | Up to day 180
  Fecal calprotectin will be reported in microgram per gram (µg/g)

SECONDARY OUTCOMES:
Changes in serum liver function tests | Up to day 180
  Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), and Alkaline Phosphatase (ALKP) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Nadeem Aslam, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslam MN, McClintock SD, Attili D, Pandya S, Rehman H, Nadeem DM, Jawad-Makki MAH, Rizvi AH, Berner MM, Dame MK, Turgeon DK, Varani J. Ulcerative Colitis-Derived Colonoid Culture: A Multi-Mineral-Approach to Improve Barrier Protein Expression. Front Cell Dev Biol. 2020 Nov 23;8:577221. doi: 10.3389/fcell.2020.577221. eCollection 2020. PMID 33330453
- [Background] Attili D, McClintock SD, Rizvi AH, Pandya S, Rehman H, Nadeem DM, Richter A, Thomas D, Dame MK, Turgeon DK, Varani J, Aslam MN. Calcium-induced differentiation in normal human colonoid cultures: Cell-cell / cell-matrix adhesion, barrier formation and tissue integrity. PLoS One. 2019 Apr 17;14(4):e0215122. doi: 10.1371/journal.pone.0215122. eCollection 2019. PMID 30995271
- [Background] McClintock SD, Attili D, Dame MK, Richter A, Silvestri SS, Berner MM, Bohm MS, Karpoff K, McCarthy CL, Spence JR, Varani J, Aslam MN. Differentiation of human colon tissue in culture: Effects of calcium on trans-epithelial electrical resistance and tissue cohesive properties. PLoS One. 2020 Mar 5;15(3):e0222058. doi: 10.1371/journal.pone.0222058. eCollection 2020. PMID 32134920
- [Background] Aslam MN, Bassis CM, Bergin IL, Knuver K, Zick SM, Sen A, Turgeon DK, Varani J. A Calcium-Rich Multimineral Intervention to Modulate Colonic Microbial Communities and Metabolomic Profiles in Humans: Results from a 90-Day Trial. Cancer Prev Res (Phila). 2020 Jan;13(1):101-116. doi: 10.1158/1940-6207.CAPR-19-0325. Epub 2019 Nov 26. PMID 31771942
- [Background] Aslam MN, McClintock SD, Jawad-Makki MAH, Knuver K, Ahmad HM, Basrur V, Bergin IL, Zick SM, Sen A, Turgeon DK, Varani J. A Multi-Mineral Intervention to Modulate Colonic Mucosal Protein Profile: Results from a 90-Day Trial in Human Subjects. Nutrients. 2021 Mar 14;13(3):939. doi: 10.3390/nu13030939. PMID 33799486
- [Background] Varani J, McClintock SD, Aslam MN. Organoid culture to study epithelial cell differentiation and barrier formation in the colon: bridging the gap between monolayer cell culture and human subject research. In Vitro Cell Dev Biol Anim. 2021 Feb;57(2):174-190. doi: 10.1007/s11626-020-00534-6. Epub 2021 Jan 5. PMID 33403624
- [Background] Varani J, McClintock SD, Aslam MN. Cell-Matrix Interactions Contribute to Barrier Function in Human Colon Organoids. Front Med (Lausanne). 2022 Mar 10;9:838975. doi: 10.3389/fmed.2022.838975. eCollection 2022. PMID 35360746
- [Derived] Aslam MN, Turgeon DK, Appelman HD, Stidham R, McClintock S, Allen R, Moraga G, Harber I, Jencks KJ, McNeely MM, Sen A, Jepsen KJ, Varani J. A multi-mineral intervention to improve disease-related and mechanistic biomarkers in ulcerative colitis patients: Results from a randomized trial. PLoS One. 2025 Dec 8;20(12):e0337408. doi: 10.1371/journal.pone.0337408. eCollection 2025. PMID 41359652